CLINICAL TRIAL: NCT00531128
Title: A Nutrigenomics Intervention for the Study of the Role of Dietary Sitosterol on Lipid, Glucose and Energy Metabolism
Brief Title: The Effect of Dietary Sitosterol on Blood Sugar and Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Prevention
Other Study IDs: 070219; 07-DK-0219
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05-17

CONDITIONS: Sitosterolemia
Keywords: Sitosterol; Nutrigenomics; Gene Expression; Insulin Resistance; Sitosterolemia
MeSH Terms: conditions — Sitosterolemia; Insulin Resistance

INTERVENTIONS:
Behavioral: High/Low Sitosterol

SUMMARY:
This study will determine if dietary supplements of sitosterol (a plant cholesterol commonly found in vegetables) can modify blood sugar and cholesterol levels and reduce the stiffness of the blood vessels in people with an abnormal copy of a gene that causes sitosterolemia. People who carry only one copy of the abnormal gene are healthy but have increased blood levels of sitosterol. People with two abnormal copies of the gene have increased levels of sitosterol and have an increased risk of heart attack. This condition is called sitosterolemia. Although extremely rare in the general population, up to 4% of the Amish carry an abnormal copy of this gene.

People of Amish background who are 18 years of age or older and in whom one person carries one copy of the abnormal gene that causes sitosterolemia and the other does not have an abnormal gene may be eligible for this study. Subjects must be of the same sex and within 5 years of age of each other.

During two periods of one month each participants receive pills containing sitosterol and then a special diet and meal supplements to change the levels of sitosterol in the diet. During only one of the two study periods, subjects receive sitosterol supplements in the pills for one month and then for 10 days in the diet. At the end of each study period, subjects come to the NIH Clinical Center for one day for the following tests:

* Measurements of height, weight, blood pressure and heart rate.
* Adipose (fat) tissue biopsy. A small piece of fat from under the skin of the abdomen is removed to examine how sitosterol affects fat tissue and its ability to process sugar and fat.
* Indirect calorimetry. A plastic transparent hood is placed over the subject s head to collect the air that is breathed for about one-half hour to study how the body uses sugar to generate energy.
* Endothelial vascular function. An ultrasound picture of a blood vessel in the forearm is taken and a blood pressure cuff is inflated around the arm to measure the vessel s ability to stretch.
* Intravenous glucose tolerance test: A small plastic tube is placed in a vein in each arm. Then over one minute the subject receives glucose through one of the tubes. Twenty minutes later the subject is given a small amount of insulin through the same tube. Blood samples are drawn through the tube in the other arm at frequent intervals for 3 hours. This test measures how sitosterol affects how the body processes sugar.
* DEXA scan. The subject lies on an x-ray table for 20 minutes during the scan, which measures total body fat.

DETAILED DESCRIPTION:
The relative distribution of the various amounts of lipids in the membranes of the adipocytes plays an important role in lipid metabolism and energy homeostasis. Sitosterolemia, a rare genetic disease is caused by a defective ABC transporter in the gut and biliary tract, which results in increased absorption and decreased excretion of plant sterols, ultimately leading to accelerated atherosclerosis and premature death.

Very recently, a mutation of the ABCG8 gene, very rare in the general population, has been described in 4% of the Old Order Amish, a well-characterized founder population in Lancaster County, Pennsylvania. Preliminary data indicate that otherwise healthy carriers (heterozygotes) of the mutation showed, as compared to controls, reduced body mass index, more large buoyant LDL cholesterol, decreased carotid intima media thickness (IMT), and a trend toward lower insulin and glucose levels, consistent with an improved metabolic syndrome profile. These data suggest that a mild excess in plant sterols could play a role in the modulation of the energy metabolism, and that dietary sitosterol may improve lipid profile and other aspects of the metabolic syndrome in genetically normal subjects.

In order to characterize mechanistically the effects of sitosterol, the most abundant plant sterol in the diet, on the development of the metabolic syndrome, we propose to study in greater detail the carriers of the ABCG8 gene mutation; that will provide the opportunity to analyze new insights into dietary sitosterol and its role in lipid and energy metabolism. We hypothesize that sitosterol in the diet will affect metabolic syndrome indices differentially in carriers of the mutation as compared to non-carriers.

We will perform a nutrigenomics intervention on 15 ABCG8 mutation carriers and sex-matched unaffected persons (age +/- 5 years). They will be treated with high-, low- sitosterol iso-caloric diets. Study subjects will be then evaluated in the NIH Clinical Center for changes in the following parameters: circulating lipids and free fatty acids, glucose disposal, resting energy expenditure and RQ, and endothelial vascular function. The Division of Endocrinology, Diabetes and Nutrition at the University Of Maryland School of Medicine will carry out the genotyping, study volunteer recruitment, cell membrane lipid content analysis, and ex-vivo adipocyte analysis.

We hypothesize that carriers of the ABCG8 gene mutation will further improve metabolic syndrome indices when challenged with a high-sitosterol diet, and will regress toward the non-carrier controls when treated with a low-sitosterol diet. Non-carrier controls will remain unchanged or show modest improvement in metabolic syndrome indices when challenged with a high-sitosterol diet, which will worsen, compared to baseline and carrier sibs, when treated with a low-sitosterol diet.

These clinical data, combined with the in vitro analysis of the effects of sitosterol on cell membranes and adipocyte metabolism will advance knowledge in the field of lipid metabolism on the relation of lipid composition to common disorders such as the metabolic syndrome. Data obtained from this project could then potentially be translated into nutritional and therapeutic interventions in the general population.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years, male or female
* Genotype ABCG8: G574 (case) or R574 (control)
* Amish ethnicity (as self-described and from the Fisher's Book)
* Informed consent (obtained in the presence of the Amish Liaison nurse)
* Control person: same sex and age +/- 5 years from case

EXCLUSION CRITERIA:

* BMI greater than or equal to 40 kg/m(2)
* History or symptoms compatible with cardiovascular disease, including hypertension greater than or equal to 140/90 mm Hg or current therapy for hypertension or cardiovascular disease
* Allergy to lidocaine, acetaminophen with codeine, oxycodone.
* Pregnancy
* Breastfeeding
* Use of hormonal contraceptives or estrogen replacement therapy
* Diabetes mellitus, either type 1 or 2
* Hypercholesterolemia (serum levels greater than or equal to 240 mg/dL), and/or use of antilipemic therapy
* Liver disease or ALT serum level greater than two fold the upper laboratory reference limit
* Renal insufficiency or estimated creatinine clearance less than or equal to 50 mL/min
* Use of medications/dietary supplements/alternative therapies known or thought to alter lipid or carbohydrate metabolism (e.g. omega-3 fatty acids, chromium, vanadate) during the study
* Current history or symptoms compatible with psychosis including major depression (including history of hospitalization for depression, history of attempted suicide, history of suicidal ideation), and/or use of antipsychotic medications
* History of drug or alcohol abuse within the last 5 years; current use of drugs or alcohol (CAGE greater than 3)
* Keloid formation (relative to subcutaneous adipose tissue biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-09-10; Primary Completion 2012-07-27 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Circulating lipids, glucose disposal, energy expenditure.

SECONDARY OUTCOMES:
Endothelial vascular function, adipose tissue gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Maryland Amish Research, Lancaster, Pennsylvania

REFERENCES:
- [Background] Luan J, Browne PO, Harding AH, Halsall DJ, O'Rahilly S, Chatterjee VK, Wareham NJ. Evidence for gene-nutrient interaction at the PPARgamma locus. Diabetes. 2001 Mar;50(3):686-9. doi: 10.2337/diabetes.50.3.686. PMID 11246892
- [Background] Dugail I, Le Lay S, Varret M, Le Liepvre X, Dagher G, Ferre P. New insights into how adipocytes sense their triglyceride stores. Is cholesterol a signal? Horm Metab Res. 2003 Apr;35(4):204-10. doi: 10.1055/s-2003-39475. PMID 12778362
- [Background] von Bergmann K, Sudhop T, Lutjohann D. Cholesterol and plant sterol absorption: recent insights. Am J Cardiol. 2005 Jul 4;96(1A):10D-14D. doi: 10.1016/j.amjcard.2005.03.014. PMID 15992510